CLINICAL TRIAL: NCT01068535
Title: Early Vascular Wall Changes by MRI in Metabolic Syndrome vs. Metabolically Normal Pre-Menopausal Women: A Pilot Study
Brief Title: Early Vascular Wall Changes by Magnetic Resonance Imaging (MRI) in Metabolic Syndrome Versus Metabolically Normal Pre-Menopausal Women: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 35352-A
Record Dates: First submitted 2010-02-11; First posted 2010-02-15 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; MetS; premenopausal women; vascular risk; atherosclerosis detection
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lipids, LDL-Buoyancy, Apo-B, Apo-A1 Inflammatory markers: hs-CRP, SAA, IL-6, & TNF-α Vascular Adhesion Markers: VCAM, sICAM
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with Metabolic Syndrome: Pre-menopausal women with Metabolic Syndrome
  Age 35-50 and any 3 of the following:
  Fasting triglycerides ≥ 150 mg/dL, Waist measurement ≥ 35 inches, HDL < 50mg/dL, Fasting glucose ≥ 100mg/dL but <126mg/dL or Blood pressure ≥ 130/85 or taking medication to treat high blood pressure.
- Non-Metabolic Syndrome (healthy) women: Non-Metabolic syndrome pre-menopausal women age 35-50
  * Body Mass Index ≤ 25
  * Regular menstrual cycles (occur every 24-35 days)
  * Fasting glucose < 100mg/dL
  * HDL-C ≥ 50mg/dL
  * Waist measurement ≤ 35 inches
  * Fasting triglycerides < 150mg/dL

SUMMARY:
The purpose of this study is to compare the vascular permeability of blood vessel walls (of the carotid artery) in pre-menopausal women who have metabolic syndrome (syndrome of having at least 3/5 following features- increased abdominal fat, low good cholesterol (HDL-C), elevated fasting blood fats (triglycerides), elevated blood pressure, an elevated fasting glucose) versus those women who are normal weight and with normal cholesterol, blood fats, blood pressure, and blood sugar. We are using a novel technology to measure vascular permeability known as dynamic contrast enhancement magnetic resonance imaging (DCE-MRI). The primary variable is ktrans ratio which is a mathematically derived quantity obtained from DCE-MRI. We are trying to identify novel markers of early atherosclerosis in young women.

DETAILED DESCRIPTION:
This study involves a phone screen & 2 study visits:

* Screening visit, which includes a quick finger stick cholesterol, glucose, triglycerides test (cholestech) to determine qualification, waist measurement, weight. Results are provided regardless of qualification. If the volunteer qualifies, a full blood draw (approximately 45cc or 3 Tablespoons) will occur. A snack is provided once blood is drawn. Additional study visit procedures include a medical history questionnaire including menstrual history, height & weight measurement, vital signs, and waist & hip measurements. This study lasts up to 90 minutes.
* MRI visit (to occur within a week of screening visit) occurs once serum pregnancy & creatinine results are received & only if approved to continue by P.I. (e.g. negative serum pregnancy and eGFR>60). An IV catheter is placed in the antecubital vein to administer an injection of (gadolinium) contrast medium. A coil is placed on each side of the subject's neck while laying flat on a bench, with her upper body inside the MRI scanner. The entire MRI procedure takes approximately 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women (age 35-50)

  * still having menstrual periods

Exclusion Criteria:

* History of diabetes mellitus
* History of cardiovascular disease (peripheral vascular disease, coronary artery disease, cerebrovascular disease)
* Serum creatinine >1.2 mg/dL (eGFR <60 ml/min.)
* Active rheumatologic disease
* Use of hormonal contraception*
* Pregnant or planning a pregnancy within the next 3 months
* Fasting triglycerides ≥ 500 mg/dL
* Fasting LDL-C ≥ 190 mg/dL
* Currently taking lipid lowering medications*
* Currently taking vaso-active (blood pressure) medications*
* Hypertension: SBP ≥ 140 and or DBP ≥90 mm Hg
* Chronic use of aspirin (prn use is allowed)
* Chronic use of non-steroidal anti-inflammatory medications (prn use is allowed)
* Tobacco use within 3 months of starting study
* Participation in another clinical trial within the last 30 days
* MRI specific exclusion criteria:

  * History of claustrophobia
  * History of decrease in kidney function (eGFR <60 ml/min.)
  * History of reaction to a contrast medium or dye used for an MRI, CT Scan, or X-ray
  * History of significant anemia or other blood disease
  * History of seizures
  * MRI-incompatible metal such as internal metal hardware or devices * Drugs within the following classifications are exclusionary: Antilipemics, antilipidemics, beta blockers, ACE inhibitors, angiotensin receptor blockers, diuretics, calcium channel blockers, alpha blockers, nitrates, and all hormonal contraceptives

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre-menopausal Women
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
ktrans of the carotid artery wall | baseline
  Ktrans is a transfer constant that is a measure of vascular permeability.

SECONDARY OUTCOMES:
carotid artery intima-media thickness as measured by MRI | baseline
  Carotid intima-media thickness is a measure of the actual thickness of the intima and media layers of the carotid artery wall.

CONTACTS AND LOCATIONS:
Overall Officials: Pathmaja Paramsothy, M.D.,M.S., Principal Investigator — University of Washington
Locations (1):
- Harborview/University of Washington, Seattle, Washington, United States